CLINICAL TRIAL: NCT00609570
Title: Effects of Nutritional Supplements on Blood Pressure and Heart Rate Variability
Brief Title: Nutritional Supplements on Blood Pressure 2008
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Logan College of Chiropractic (Other)
Responsible Party: John Zhang, Logan University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: RD0920070111
Record Dates: First submitted 2008-01-25; First posted 2008-02-07 (Estimated); Last update posted 2008-10-28 (Estimated); Status verified 2008-10

CONDITIONS: Hypertension
Keywords: hypertension; supplement; HRV
MeSH Terms: conditions — Hypertension | interventions — Whey Proteins

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Fruit and vegetables (Experimental): Fruits and vegetables
  Interventions: Dietary Supplement: NanoGreens
- Whey protein (Active Comparator): Whey protein
  Interventions: Dietary Supplement: Whey protein
- Ca (Active Comparator): Calcium pills
  Interventions: Dietary Supplement: Calcium pills

INTERVENTIONS:
Dietary Supplement: NanoGreens — fruits and vegetables
  Arms: Fruit and vegetables
Dietary Supplement: Whey protein — Whey
  Other Names: NanoPro
  Arms: Whey protein
Dietary Supplement: Calcium pills — CA
  Other Names: CA
  Arms: Ca

SUMMARY:
Three different supplements will be used in the study (fruits and vegetable powders, whey protein and calcium) for patients with hypertension. The null hypothesis was that the supplements had no effects on participants' blood pressure.

DETAILED DESCRIPTION:
Hypertensive participants will be randomly assigned into three groups. The first group of participants will take the fruits and vegetable powders mixed with water. The second group takes whey protein and the third group takes calcium pills. Blood pressure and heart rate variability will be measured every two weeks for three months.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-70
* Hypertensive male and female subjects.

Exclusion Criteria:

* Severe cardiovascular and renal conditions.
* Pregnancies and taking medications.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-07 (Estimated); Study Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
Blood pressure and HRV | every two weeks for three months

CONTACTS AND LOCATIONS:
Overall Officials: John Zhang, MD, PhD, Study Chair — Logan University
Locations (2):
- United States (2):
  - Logan University, College of Chiropractic, Chesterfield, Missouri
  - Logan University, Chesterfield, Missouri